CLINICAL TRIAL: NCT03925623
Title: Design Factors for Evaluating Child Resistant Packaging
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Laura Bix, Professor, Michigan State University
Other Study IDs: MSU17-1447
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Unintentional Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Commercial closure system: Participants (42-54 months of age) will be assigned to try to open one of three treatments. One cohort will receive a 38/400 bottle equipped with a standard two piece push and turn cap and asked to open this during 2 five minute trials.
  Interventions: Other: Novel approaches for the design of child resistant closures
- Physically based design strategy: Participants (42-54 months of age) will be assigned to try to open one of three treatments. One cohort will receive a 38/400 bottle equipped a novel closure that was designed using anthropometric data such that it disallows children from engaging the system and enables adults. Children will be asked to open this during 2 five minute trials.
  Interventions: Other: Novel approaches for the design of child resistant closures
- Cognitively based design strategy: Participants (42-54 months of age) will be assigned to try to open one of three treatments. One cohort will receive a 38/400 bottle equipped with the design feature that was introduced as part of the physical intervention (above); however, this treatment is sized such that children should be able to engage it (if they understand how). In having these three treatments, we began to evaluate the paradigm which enables the design to work. (Do they fail to understand how?- Cognitive treatment fail- and or Can they not effectively manipulate the closure? --- Physical failure).
  Interventions: Other: Novel approaches for the design of child resistant closures

INTERVENTIONS:
Other: Novel approaches for the design of child resistant closures — Two novel designs for child resistant closures are tested.
  One is sized based on the anthropometric properties of adults and children's hands such that it should disallow children from engaging the system and enable adults (the physically based design strategy). The other replicates the first design, but is sized such that either of the two populations should be able to engage the closure.
  In testing this way, we begin to differentiate the paradigm that holds the children out (the cognitively based design strategy-- they do not understand and/or a physical one- they are unable to use the closure).
  Results (proportion of children opening within the first or second five minute periods of test and time to opening during the same) from each of these, will be compared to results from the third treatment, a standard, commercially available push and turn system.

SUMMARY:
Each year over 59,000 children under the age of 5 are taken to emergency rooms (equivalent to 4 busloads of children arriving every day to the ER) because they were able to get into medication containers unsupervised. 95 percent of these ER visits occurred due to the child getting into medicine when an adult was not looking.

Child resistant containers (CRC) are intended to restrict entry by imposing a cognitive barrier (the child must understand how to operate the CRC mechanism in order to open it) and a physical barrier (the child must posses the motor skills necessary to operate the CRC).

Investigators are testing a design which changes the physical area available for grip utilizing anthropometric data that, in theory, would exclude children and enable adults.

Investigators will evaluate the proposed design's effectiveness in two ways (1: cognitive barrier) will the child understand where they need to specifically grip the cap with their fingers and (2: physical barrier) will the child be able to use an appropriate gripping strategy to apply enough torque to rotate the cap and open it.

DETAILED DESCRIPTION:
In order to evaluate the effectiveness of cognitive and physical barriers as child resistant design features, investigators are testing designs which change the physical area available for grip utilizing anthropometric data that, in theory, would exclude children and enable adults. Testing will be conducted with children aged between 42-54 months of age. Our testing is adapted from testing dictated by 16 CFR 1700; this testing is mandated by the Poison Prevention Packaging Act of 1970 and is used throughout the United States (and, in fact, adapted by much of the world) to verify the performance of child resistant packaging. The maximum age limit specified by 16 CFR 1700 is 51 months so the child testing for this study represents a more severe test of the closure.

One type of package is being tested: a 38mm diameter neck 400 thread finish (38/400) bottle that is typical of what is used to hold over-the-counter (OTC) medications. The bottle is outfitted with a two-piece continuous thread screw cap closure. Three treatments of the screw cap are being evaluated. One treatment attempts to restrict children from accessing the package using a cognitive paradigm (design intuitiveness for opening) the second treatment leverages a physical paradigm (anthropometric characteristics of the hand to keep them out) and the third treatment, the control, is a standard OTC push-down and turn child resistant screw cap.

Summary

Children will be recruited with the help of the Michigan State University Child Development Labs (MSU CDL) and testing will take place in a designated room within the Wilkshire Early Childhood Center in Haslett, Michigan and/or Early Learning Institute (ELI) preschool in East Lansing, MI. Approximately 120 children will test a single treatment of the three (N=40 per treatment); attempts will be made to counterbalance age and sex by treatment . The width of each child's thumbs will be measured by taking a digital photographic with their hand place on a grid of known dimensions. Testing will then occur in two 5 minute segments for each treatment (as with the regulated protocol overseen by CPSC).

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 42 months to 54 months at the time of testing Have IRB approved consent form signed by parent or guardian Haver permission to be video taped Provide verbal assent (or assent through body language- head nod, etc)

Exclusion Criteria:

* No history of food allergies of any kind
* No known issues with lactose, including lactose intolerance or allergy
* Have no physical or mental impairments that impact their ability to open packages

Ages: 42 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 42-54 months of age Recruited from preschools throughout mid Michigan
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Proportion of successful openings within a given treatment | First five minutes OR Second five minutes
  Openings are recorded in binary fashion (child was successful yes/no)
Time to successful opening | First five minutes OR Second five minutes
  The time it took for children to successfully open the packaging

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Michigan State University Child Development Laboratory- East Lansing, East Lansing, Michigan
  - School of Packaging, East Lansing, Michigan
  - Wilkshire Early Childhood Center-, Haslett, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Raw flat file will be available deidentified. Not even the research team will be able to tie data to subject identity
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2019
Access Criteria: Will be provided with publications as a deidentified flat file as required by editors